CLINICAL TRIAL: NCT07260760
Title: Clinical Comprehensive Evaluation of Neuroprotective Drugs for Acute Ischemic Stroke
Acronym: Ischemic strok
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, LI YAN, Chief Pharmacist, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2025(206)
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Neuroprotective drugs; Real-world studies
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study conducted a comprehensive evaluation of commonly used neuroprotective agents in acute ischemic stroke, assessing their real-world value across six dimensions: safety, efficacy, cost-effectiveness, innovativeness, appropriateness, and accessibility. Employing a prospective observational design, it primarily investigates the association of edaravone and dexrazoxane with clinical outcomes in patients with mild-to-moderate stroke, with subgroup analyses performed according to Trial of Org 10172 in Acute Stroke Treatment （TOAST ）classification.

DETAILED DESCRIPTION:
A comprehensive evaluation of commonly used clinical neuroprotective drugs was conducted, analyzing their practical application value in acute ischemic stroke treatment across six dimensions: safety, efficacy, cost-effectiveness, innovation, appropriateness, and accessibility. In a real-world clinical setting, this prospective observational study design primarily evaluates the association between edaravone and dexrazoxane usage and the efficacy and safety outcomes in patients with mild-to-moderate ischemic stroke, while conducting subgroup analyses based on different Trial of Org 10172 in Acute Stroke Treatment （TOAST ）classifications.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age≥18

  2: Acute ischemic stroke in the anterior circulation occurring within 48 hours

  3: Baseline NIHSS score of 1-15 points (mild stroke: baseline NIHSS score of 1-5 points; moderate stroke: baseline NIHSS score of 6-15 points)

  4: Pre-onset mRS score≤1

  5: Use of Edaravone (injection or tablets)

  6: Exclude intracranial hemorrhage

  7: Sign the informed consent form

Exclusion Criteria:

* 1: A head CT or MRI scan indicates the presence of intracranial hemorrhagic disease

  2: Patients with cerebral embolism or suspected cerebral embolism who also have severe atrioventricular block, atrial fibrillation, myocardial infarction, valvular heart disease, infective endocarditis, or a heart rate below 50 beats per minute

  3: Abnormal liver function (ALT or AST transaminase levels exceeding the upper limit of normal), abnormal kidney function (creatinine levels exceeding the upper limit of normal), or individuals with other severe systemic diseases, etc

  4: Allergy to the test drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale（mRS ）scores of 0-1 | 90 days

SECONDARY OUTCOMES:
Proportion of patients with mRS scores of 0-2 | 30 days
Percentage reduction in National Institutes of Health Stroke Scale （NIHSS ）score compared to pre-treatment | 90 days after medication

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofang Niu, Principal Investigator — Heze Municipal Hospital; Leqing Zhang, Principal Investigator — Yanggu County People's Hospital; Lei Duan, Principal Investigator — Zibo Central Hospital; Kai Ren, Principal Investigator — Haiyang People's Hospital; Rongrong Zhang, Principal Investigator — Sishui County People's Hospital; Ping Yang, Principal Investigator — Jinan Fourth People's Hospital; Ning Liu, Principal Investigator — Shandong Hospital of Integrated Traditional Chinese and Western Medicine; Pengcheng Du, Principal Investigator — Qilu Hospital of Shandong University, Dezhou Branch; Hui Liu, Principal Investigator — Jinan Municipal People's Hospital; Xi Rong, Principal Investigator — Weifang Yidu Central Hospital; Deyin Zhai, Principal Investigator — Linyi Traditional Chinese Medicine Hospital; Zhiqiang Zhang, Principal Investigator — Anqiu People's Hospital; Jiyong Wu, Principal Investigator — Shandong Provincial Second People's Hospital; Meixia Wang, Principal Investigator — Jining Medical University Affiliated Hospital; Ping Wang, Principal Investigator — Liaocheng People's Hospital; Jiyao Li, Principal Investigator — Liaocheng Municipal People's Hospital

REFERENCES:
- [Result] Fu Y, Wang A, Tang R, Li S, Tian X, Xia X, Ren J, Yang S, Chen R, Zhu S, Feng X, Yao J, Wei Y, Dong X, Ling Y, Yi F, Deng Q, Guo C, Sui Y, Han S, Wen G, Li C, Dong A, Sun X, Wang Z, Shi X, Liu B, Fan D. Sublingual Edaravone Dexborneol for the Treatment of Acute Ischemic Stroke: The TASTE-SL Randomized Clinical Trial. JAMA Neurol. 2024 Feb 19;81(4):319-26. doi: 10.1001/jamaneurol.2023.5716. Online ahead of print. PMID 38372981